CLINICAL TRIAL: NCT04838197
Title: Understanding Caregiver Burden When Traditional Total Hip and Knee Replacement Surgeries Shift From Inpatient Hospitalization to Outpatient Settings: A Prospective Cohort Study
Brief Title: Understanding Caregiver Burden for Hip and Knee Replacement Surgery Patients
Status: Completed | Type: Observational
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0045-E
Record Dates: First submitted 2021-03-30; First posted 2021-04-09 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Caregiver Burnout
Keywords: Total Joint surgeries; Total Knee Arthoplasty; Total Hip Arthoplasty
MeSH Terms: conditions — Caregiver Burden | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregiver: If the caregiver agrees and consents to participating in the study, basic demographic and social data will be collected at baseline. The caregiver will also complete the caregiver burden questionnaire via telephone call at five different time points: pre-operatively, and post-operative 48 hours, 1 week, 2 weeks, and 1 month.
  Interventions: Other: Questionnaires and Surveys

INTERVENTIONS:
Other: Questionnaires and Surveys — Quantitative questionnaires will measure and quantify the importance of the various factors (e.g., intensity of dependence, duration of care, health literacy, physical well-being, emotional well-being, social well-being, and financial well-being) that contribute to caregiver burden both preoperatively and postoperatively at 48 hours, 1 week, 2 weeks, and 1 month.

SUMMARY:
Caregiver burden is the response to the emotional, financial, physical, psychological, and social stressors associated with having to care for another family member. Previous studies have looked at the impact of caregiver burden in caregivers caring for loved ones dealing with long-term disease, such as dementia. The research has found that one in three caregivers suffer from depression, and experience high levels of stress and anxiety. However, these findings may not be relatable to the outpatient surgical setting. The purpose of this study is to find out how various factors such as the physical, emotional, social, and financial burden impact caregivers who are responsible for providing care to patients who are undergoing same-day surgical procedures that are traditionally performed as inpatient surgery. By understanding this potential burden on the caregiver, we hope that future healthcare improvements can be made to minimize this impact on the patients and their caregiver.

DETAILED DESCRIPTION:
The extent of caregiver burden in the acute postoperative outpatient settings, immediately following major orthopedic surgery that has traditionally been performed in an inpatient setting, remains unknown. Care giving places a tremendous amount of physical and mental stress onto the caregiver, which may result in the "hidden patient" in the caregiver. It is expected that by 2026, 51% of TJA will be performed as outpatient procedures. Building on the successes of the country's first outpatient TKA program at Women's College Hospital, and with the expansion to include outpatient THA procedures, it is now important to understand whether or not our innovative ambulatory model is simply transferring the burden of postoperative care and recovery from nurses, doctors, and other hospital staff to family members, friends, or privately-employed caregivers.

In the current state of literature, there is inadequate data examining caregiver burden when traditional surgical procedures are shifted to an outpatient setting, therefore, a comprehensive study is required to understand the various dimensions of caregiver burden. Therefore, our research question is "what are the most important factors that contribute to the burden of care for caregivers of patients undergoing outpatient surgical procedures traditionally performed as inpatients?"

This prospective cohort study examines how the various dimensions of caregiver burden impact caregivers at different time points throughout the care giving experience. These dimensions include factors such as the intensity of dependence on the caregiver, duration of care, caregiver specific factors (e.g., the health literacy of the caregiver), and care giving dimensions (e.g., physical, emotional, social and financial burdens). Through gaining an understanding of how the various dimensions of caregiver burden impact caregivers in the outpatient settings, meaningful improvements can be made in the future and ultimately improve the quality of life of the caregiver during the time of care.

ELIGIBILITY:
Inclusion Criteria (Patient):

* Undergoing ambulatory total knee or total hip arthroplasty
* Patient is able to consent for self

Inclusion Criteria (Caregiver):

* English speaking, or willing to use an interpreter
* Over the age of 18 years
* Primarily responsible for providing care to the patient undergoing ambulatory total knee or total hip arthroplasty

Exclusion Criteria (Patient and Caregiver):

* Refusal or unable to provide informed consent
* The patient is a resident in a nursing home or is already receiving daily professional care for most ADLs
* Unable to complete data collection tools or take part in telephone interviews due to cognitive or physical impairment

Withdrawal Criteria After Enrollment

* Patient or Caregiver refusal to participate or continue with the study at any point
* Cancellation of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing ambulatory TKA or THA will be approached for consent. Their primary caregivers will be consented to participate as well.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Care-giver experience assessment with homegrown quantitative questionnaires | before surgery up to discharge, assessed up to 1 month
  To gain an understanding of the various factors contributing to the burden of care experienced in the post-operative setting among our caregivers caring for patients undergoing TKA or THA within our ambulatory model.
  (e.g., intensity of dependence, duration of care, health literacy, physical well-being, emotional well-being, social well-being, and financial well-being) On a scale of 5-Point Likert Scale from Strongly Disagree to Strongly Agree

SECONDARY OUTCOMES:
Intensity of patient dependence on the caregiver | at 48 hours, 1 week, 2 weeks, and 1 month post-operatively
  Using the Katz Index of Independence in Activities of Daily Living
Time expected to care for the patient | at 48 hours, 1 week, 2 weeks, and 1 month post-operatively
  This section will ask caregivers about the number of hours they spend/expect to spend performing caregiving activities.
Number of people the caregiving responsibilities have been shared with | at 48 hours, 1 week, 2 weeks, and 1 month post-operatively
  This section will ask caregivers questions focusing on their health literacy, defined as "the ability to obtain, read, understand and use healthcare information". Caregivers will be asked how prepared/confident they feel performing the necessary medical caregiving tasks, and if they have sought out additional medical information from healthcare professionals, or online resources to help assist in a caregiving task. Finally, caregivers will be asked to identify if they have shared the caregiving responsibilities with another person throughout the caregiving experience
Caregivers' preparedness | at 48 hours, 1 week, 2 weeks, and 1 month post-operatively
  This section will ask caregivers questions focusing on their health literacy, defined as "the ability to obtain, read, understand and use healthcare information". Caregivers will be asked how prepared/confident they feel performing the necessary medical caregiving tasks, and if they have sought out additional medical information from healthcare professionals, or online resources to help assist in a caregiving task. Finally, caregivers will be asked to identify if they have shared the caregiving responsibilities with another person throughout the caregiving experience
Caregivers' reliance on additional medical information to help assist in care-giving | at 48 hours, 1 week, 2 weeks, and 1 month post-operatively
  This section will ask caregivers questions focusing on their health literacy, defined as "the ability to obtain, read, understand and use healthcare information". Caregivers will be asked how prepared/confident they feel performing the necessary medical caregiving tasks, and if they have sought out additional medical information from healthcare professionals, or online resources to help assist in a caregiving task. Finally, caregivers will be asked to identify if they have shared the caregiving responsibilities with another person throughout the caregiving experience
Caregivers' perceptions on the physical demands of caregiving | pre-operatively and post-operatively at 48 hours, 1 week, 2 weeks, and 1 month
  This section will ask caregivers questions regarding the impact of caregiving on their physical well-being. Caregivers will be asked pre-operatively if they expect caring for the patient will be physically demanding, and post-operatively if caring for the patient has been physically demanding. As well, caregivers will be asked if preparing for/caring for the patient has disrupted their sleep
Disruption to the caregivers sleep | pre-operatively and post-operatively at 48 hours, 1 week, 2 weeks, and 1 month
  This section will ask caregivers questions regarding the impact of caregiving on their physical well-being. Caregivers will be asked pre-operatively if they expect caring for the patient will be physically demanding, and post-operatively if caring for the patient has been physically demanding. As well, caregivers will be asked if preparing for/caring for the patient has disrupted their sleep
Presence of depression and anxiety within caregivers | pre-operatively and post-operatively at 48 hours, 1 week, 2 weeks, and 1 month
  To further measure anxiety and depression, caregivers will complete the Hospital Anxiety and Depression Scale (HADS). HADS was designed to be a reliable, valid, and simple to use tool to identify and quantify anxiety and depression. Though the term 'hospital' in the title suggests it only valid in the hospital setting, many studies have confirmed the tools valid use in primary care medical and community settings. HADS is comprised of 14 items, 7 assessing anxiety and 7 assessing depression.
Disruption to the caregivers' emotional well-being | pre-operatively and post-operatively at 48 hours, 1 week, 2 weeks, and 1 month
  This section will ask caregivers questions regarding the impact of caregiving on their emotional well-being. Caregivers will be asked if preparing for/caring for the patient has disrupted their emotional well-being (e.g., anxious, depressed, irritable, angry, etc.).Each item is rated on a 4-point scale ranging from 0 meaning no not at all, to 3 meaning yes definitely. The total score for each sub scale ranges from 0-21, where 0-7 indicates non-cases, 8-10 indicates mild cases, 11-14 indicates moderate cases, and 15-21 indicates cases of anxiety or depression.
Disruption to the caregivers' social well-being | pre-operatively and post-operatively at 48 hours, 1 week, 2 weeks, and 1 month
  This section will ask caregivers questions regarding the impact of caregiving on their social well-being. Caregivers will be asked if preparing for/caring for the patient has disrupted their social well-being (e.g., socializing with friends and family, participating in recreational/leisure activities, etc.).
Presence of financial strain due to caregiving | pre-operatively and post-operatively at 48 hours, 1 week, 2 weeks, and 1 month
  This section will ask caregivers questions regarding the impact of caregiving on their financial health. Caregivers will be asked if preparing for/caring for the patient has caused financial strain. Caregivers will be asked to identify how many days they expect to take off work to care for the patient, and how many days they actually took off work to care for the patient. Likewise, caregivers will be asked how much out of pocket they expect to spend on the patient during the caregiving experience, and then on post-operative 1 month they will be asked how much they actually spent on the patient during the caregiving experience.
Number of days expected to be taken off work to help care for the patient | pre-operatively, and the actual number of days taken off to help care for the patient at 1 month
  This section will ask caregivers questions regarding the impact of caregiving on their financial health. Caregivers will be asked if preparing for/caring for the patient has caused financial strain. Caregivers will be asked to identify how many days they expect to take off work to care for the patient, and how many days they actually took off work to care for the patient. Likewise, caregivers will be asked how much out of pocket they expect to spend on the patient during the caregiving experience, and then on post-operative 1 month they will be asked how much they actually spent on the patient during the caregiving experience.
Amount expected to be spent throughout the caregiving experience | pre-operatively, and the amount spent during the caregiving experience at 1 month
  This section will ask caregivers to identify which factors are contributing the greatest to caregiver burden at various time points throughout the caregiving experience. Caregivers will be asked: "If you were given $1,000 to spend immediately to help ease the caregiving experience, how would you allocate your spending on the following factors?" Caregivers will be able to allocate the money among the seven factors previously mentioned, with hopes that caregivers will be allocating the money to different factors that are contributing significantly to the caregiver burden at various time points.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No